CLINICAL TRIAL: NCT07085507
Title: A Phase 1/2, Randomized, Double-Blind, Placebo-Controlled, Single and Multiple Dose Escalation Study in Healthy Participants and an Expansion Cohort in Adult Patients With Multiple Sclerosis to Characterize the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of VT7208
Brief Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of VT7208 in Healthy Participants and MS Patients
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vidya Therapeutics Inc (Industry)
Collaborators: Vidya Therapeutics Australia Pty Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VT7208-101
Record Dates: First submitted 2025-07-07; First posted 2025-07-25 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Multiple Sclerosis
Keywords: pharmacokinetics; healthy volunteers; pharmacodynamics; central nervous system
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Part 1 SAD Cohorts: Active drug (Experimental): Participants will receive a single dose of VT7208 in a dose escalation format.
  Interventions: Drug: VT7208
- Part 1 SAD Cohorts: Placebo (Placebo Comparator): Healthy volunteers will receive a single dose of placebo
  Interventions: Drug: Placebo
- Part 1 MAD Cohort: Active drug (Experimental): Healthy volunteers will receive repeated doses of VT7208. Dose to be determined based on escalation data from SAD Cohorts
  Interventions: Drug: VT7208
- Part 1 MAD Cohort: Placebo (Placebo Comparator): Healthy volunteers will receive repeated doses of placebo comparator.
  Interventions: Drug: Placebo
- Part 2: Food Effect (Experimental): Open label randomized cohort to be administered to healthy volunteers. Participants will be randomized to receive dose in either fasted or fed state. Dose to be determined from data of SAD and MAD cohorts.
  Interventions: Drug: VT7208
- Part 3: Patients with Multiple Sclerosis (Experimental): Open label cohort to be administered to patients with MS. Dose for this part will be determined from parts 1 and 2.
  Interventions: Drug: VT7208

INTERVENTIONS:
Drug: VT7208 — a small synthetic molecule capsule, oral
  Arms: Part 1 MAD Cohort: Active drug; Part 1 SAD Cohorts: Active drug; Part 2: Food Effect; Part 3: Patients with Multiple Sclerosis
Drug: Placebo — capsule, oral
  Arms: Part 1 MAD Cohort: Placebo; Part 1 SAD Cohorts: Placebo

SUMMARY:
Part 1 of this study will evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of VT7208 in healthy volunteers.

Part 2 of this study will be an open-label, randomized study to characterize the effect of food on the pharmacokinetics of VT7208 in healthy volunteers.

Part 3 of this study will evaluate the safety of VT7208 as monotherapy in patients with MS.

DETAILED DESCRIPTION:
This study is a Phase 1/2 randomized, double-blind, placebo-controlled, single- and multiple-dose study with staggered dose escalations in healthy participants.

Following completion of SAD and MAD cohorts, healthy volunteers will participate in administration of VT7208 with and without food to determine the effect of a fasted or fed state on pharmacokinetics.

Participants with MS will be recruited for part 3 of this study.

This study consists of 3 parts, as follows:

Part 1: SAD in healthy volunteers with a single dose administration of VT7208 or placebo and collection of study data.

MAD in healthy volunteers with multiple dose administration of VT7208 or placebo and collection of study data.

Part 2:

Food effect cohort in healthy volunteers. Participants will be randomized to receive open label VT7208 in either a fasted state or a fed state, and will receive the opposite at the next admission to the study site.

Part 3:

Participants MS will receive VT7208 with dose determined from Parts 1 and 2. Participation in this section will entail weekly study visits for administration of study medication collection of study data.

ELIGIBILITY:
Inclusion Criteria:

Parts 1 and 2

* Age 18-65
* Must be in good health with no significant medical history
* Willing and able to attend all study visits and comply with study requirements, including lumbar puncture for CSF collection
* Able and willing to provide written informed consent

Part 3

* Age 18-60
* Must be in good health with no significant medical history
* MS diagnosis prior to Day 1 in accordance with 2017 McDonald criteria.
* Willing and able to attend all study visits and comply with study requirements, including lumbar puncture for CSF collection
* Able and willing to provide written informed consent

Exclusion Criteria:

* Evidence of clinically significant condition or disease
* Any physical or psychological condition that prohibits study completion
* Known history of illicit drug use or drug abuse, harmful alcohol use (at the -Investigator's discretion), alcoholism, and/or smoking or nicotine-containing product use within 7 days prior to the first dose of study agent
* History of severe allergic reactions or hypersensitivity
* Donation or loss of ≥ 1 unit of whole blood or plasma within 4 weeks prior to dosing

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence, nature, and severity of treatment emergent adverse events (TEAEs) and serious adverse events (SAEs) of VT7208 in healthy volunteers and patients with MS | Up to 16 weeks
  Incidence, nature, and severity of treatment emergent adverse events (TEAEs) and serious adverse events (SAEs)

SECONDARY OUTCOMES:
Part 1: Pharmacokinetics of a single dose of VT7208 in healthy adults | up to 2 weeks
  Pharmacokinetic parameter of CMAX of VT7208 in the blood of healthy adults
Part 1: Pharmacodynamics (PD) of a single dose of VT7208 in healthy adults | up to 2 weeks
  BTK inhibition as measured by free, total and phosphorylated BTK level in blood
Part 1: Pharmacokinetics of multiple doses of VT7208 in healthy adults and in patients with MS | up to 2 weeks
  Pharmacokinetic parameter of CMAX of VT7208 in the blood of healthy adults
Part 1: Pharmacodynamics (PD) of multiple doses of VT7208 in healthy adults and in patients with MS | up to 2 weeks
  BTK inhibition as measured by free, total and phosphorylated BTK level in blood
Part 2: Pharmacokinetics of VT7208 in healthy adults fed and fasted | up to 2 weeks
  Pharmacokinetic parameter of CMAX of VT7208 in the blood
Part 2: Pharmacodynamics (PD) of VT7208 in healthy adults fed and fasted | up to 2 weeks
  BTK inhibition as measured by free, total and phosphorylated BTK level in blood of healthy adults fed and fasted
Characterize the ability of VT7208 to cross the blood brain barrier in healthy adults and in patients with MS | Up to 16 weeks
  Ability of VT7208 to cross the blood brain barrier will be measured in cerebrospinal fluid (CSF). This will be collected during admitted study visits for healthy volunteers

CONTACTS AND LOCATIONS:
Locations (1):
- CMAX, Adelaide, South Australia, Australia